CLINICAL TRIAL: NCT02436889
Title: Treatment of Incontinence Without Memory Problems
Acronym: TRIUMPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Alison Huang, MD, Associate Professor, Department of General Internal Medicne; Epidemiology & Biostatistics; Urology, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-15553
Record Dates: First submitted 2015-04-30; First posted 2015-05-07 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Urge Incontinence; Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — mirabegron; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirabegron (Experimental): Participants will be instructed to take one tablet and 1 capsule (total of 2) of blinded study medication once a day, orally, for 8 weeks. They will start with Mirabegron (25mg) dose of study medication and will have the option of dose escalation to 2 tablets and 2 capsules (total of 4) per day (Mirabegron 50mg).
  Interventions: Drug: Mirabegron
- Tolterodine Tartrate (Active Comparator): Participants will be instructed to take one tablet and 1 capsule (total of 2) of blinded study medication once a day, orally, for 8 weeks. They will start with tolterodine tartrate (4 mg) dose of study medication and will have the option of dose escalation to 2 tablets and 2 capsules (total of 4) per day tolterodine tartrate 4 mg + identical placebo.
  Interventions: Drug: Tolterodine Tartrate

INTERVENTIONS:
Drug: Mirabegron
  Other Names: Myrbetriq
  Arms: Mirabegron
Drug: Tolterodine Tartrate
  Other Names: Detrol LA
  Arms: Tolterodine Tartrate

SUMMARY:
An 8-week randomized, controlled, pilot clinical trial of Mirabegron compared to a standard anticholinergic therapy (Detrol LA) in elderly women with urgency urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling, ambulatory females ≥ 65 years old
* Urgency or Mixed Urgency Predominate Urinary Incontinence (subject-reported) for ≥ 3 months prior to Screening (Visit 1)
* On a 3-day voiding diary, documentation of at least 3 urgency incontinence episodes with the number of urgency incontinence episodes greater than number of stress incontinence episodes
* Capability of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risk and benefits
* Ability to perform all procedures and tests required by the protocol
* Report having a primary health care provider
* Willingness to remain on stable medication regime for duration of the randomized controlled trial. Participants will be asked to not add new medications during the randomized controlled trial, such as diuretics and other medications which may affect their voiding pattern.

Exclusion Criteria:

* Seated blood pressure >180/110 at Screening or Baseline
* Physician diagnosis of dementia
* Current use of dementia medications, debilitating or recent neurologic disease
* Mini Mental State Examination (MMSE) score <20
* History of urinary retention, gastric retention, uncontrolled narrow angle glaucoma, myasthenia gravis, severe ulcerative colitis, toxic megacolon, fistula or a hole in your bladder or rectum, birth defect leading to urine leakage, and urine leakage starting in childhood
* Clinically significant hepatic (Child Pugh B or greater) or renal (creatinin clearance <30 mL/min or eGFR <30 mL/min/1.73 m2)
* Neurologic conditions such as stroke, multiple sclerosis, spinal cord injury, or Parkinson's disease.
* Major cardiovascular even in the past 6 months (i.e., MI, unstable angina, hospitalization for chest pain)
* Symptomatic pelvic organ prolapse defined as participant report of feeling or seeing a bulge outside the vagina within the past 3 months.
* History of surgery for incontinence in the past 5 years, pelvic surgery the past 6 months (i.e., for prolapse or hysterectomy), intra-vesical therapy (botox), and/or bulk injections within the past 6 months.
* A known history of interstitial cystitis or a significant pain component associated with OAB symptoms, uninvestigated hematuria, urogenital cancer, radiation to the pelvis or external genitalia.
* Urinary tract infection (UTI) as shown by the results of the urinalysis at screening or recurrent urinary tract infection (RUTIs) defined as treatment for UTI >3 times in the last year.
* Urinary retention (post-void residual urine volume >150 cc measured by Bladder scan at screening.
* Use of any electrostimulation, bladder training, or pelvic floor exercises (with certified incontinence practitioners) within 4 weeks of Screening.
* Received study medication in any previous mirabegron clinical trial.
* Prior failure for either efficacy or tolerability of ≥ 2 OAB medications in the last year. (Failure: inadequate symptom control after two medications for a minimum of one month each.)
* Has been treated within 2 weeks prior to Screening and/or is currently being treated with:

  * Any drug treatment for OAB
  * Any drugs with significant anticholinergic and antispasmodic effects (see exception for tricyclic antidepressants below)
* Has started treatment with tricyclic antidepressants or estrogens within 4 weeks prior to Screening and/or is not on a stable dose.
* Intermittent use or unstable dose of diuretics. Treatment with diuretics initiated within 2 weeks prior to baseline and/or is not on a stable dose is not permitted.
* Treatment with potent CYP3A4 inhibitors, such as clarithromycin, ketoconazole, and itraconazole within 2 weeks prior to Screening.
* Administration of medications capable of inducing hepatic enzyme metabolism or transport (e.g., barbiturates, rifampicin, carbamazepine, phenytoin, primidone, or St. John's Wort) in the past 30 days.
* Administration of narrow therapeutic index drugs metabolized by CYP2D6, such as thioridazine, flecainide, and propafenone.
* Previously received any investigational drug within 30 days prior to trial entry.
* Alcohol and/or any other drug abuse in the opinion of the investigator.
* Participants who have any medical (including known history of major hematological, renal, cardiovascular, or hepatic abnormalities) or psychological condition or social circumstances that would impair their ability to participate reliably in the trial, or those who may increase the risk to themselves or others by participating.
* Participants who, in the opinion of the investigator, are not likely to complete the trial for whatever reason.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslee Subak, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirabegron: Participants will be instructed to take one tablet and 1 capsule (total of 2) of blinded study medication once a day, orally, for 8 weeks. They will start with Mirabegron (25mg) dose of study medication and will have the option of dose escalation to 2 tablets and 2 capsules (total of 4) per day (Mirabegron 50mg).
  Mirabegron
- Tolterodine Tartrate: Participants will be instructed to take one tablet and 1 capsule (total of 2) of blinded study medication once a day, orally, for 8 weeks. They will start with tolterodine tartrate (4 mg) dose of study medication and will have the option of dose escalation to 2 tablets and 2 capsules (total of 4) per day tolterodine tartrate 4 mg + identical placebo.
  Tolterodine Tartrate
Period: Overall Study
Arm/Group | Mirabegron | Tolterodine Tartrate
Started | 12 | 11
Completed | 11 | 10
Not Completed | 1 | 1
Not completed — No improvement in symptoms | 1 | 0
Not completed — Does not like/could not tolerate medicat | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirabegron | Tolterodine Tartrate | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Customized [Count of Participants; unit: Participants]
  65-69 years | 5 | 7 | 12
  70-79 years | 7 | 3 | 10
  80-89 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Asian American | 0 | 1 | 1
  American Indian/Alaska Native | 0 | 0 | 0
  African American | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White or Caucasian | 11 | 10 | 21
  Other Race | 1 | 0 | 1
  Hispanic or Latina | 1 | 0 | 1
  Not Hispanic or Latina | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23
Incontinence Frequency [Mean (Standard Deviation); unit: Episodes per day] — Urinary incontinence refers to any involuntary leakage of urine. Urge incontinence (also known as urgency incontinence) refers to involuntary leakage of urine that occurs as a result of a sudden or strong urge to urinate, when an individual cannot reach the toilet in time)
  Episodes per day
    Total Urge Incontinence | 3.87 (2.33) | 4.48 (1.92) | 4.16 (2.11)
    Total Urinary Incontinence | 4.43 (3.20) | 4.96 (1.98) | 4.68 (2.64)
California Verbal Learning Test [Mean (Standard Deviation); unit: Trials 1-5 Free Recall Total] — The California Verbal Learning Test involves the presentation of one list of 16 words taken from three categories. Following a brief delay, the participant is asked to recall the words. Memory is then tested after another 20-minute delay. Trials 1-5 free recall is the total number of correctly remembered items (for trials 1-5). This would make the possible range for this score 0-80, with a higher score being better.
  Trials 1-5 Free Recall Total | 51.36 (12.29) | 49.50 (10.98) | 50.48 (11.43)
Short Physical Performance Battery [Mean (Standard Deviation); unit: Score on Scale] — Range 0-12, higher score indicates better functioning.
  Score on Scale | 10.67 (2.1) | 11.00 (2.2) | 10.83 (2.1)
Trail Making Test [Mean (Standard Deviation); unit: seconds] — These are timed, written tests with shorter test times corresponding to better attention, visual scanning, and executive function.
  seconds
    Trail A Time (0-150 sec) | 40.33 (26.3) | 35.06 (9.5) | 37.81 (19.9)
    Trail B Time (0-300 sec) | 93.03 (61.5) | 85.39 (29.4) | 89.38 (47.9)
Instrumental Activities of Daily Living [Mean (Standard Deviation); unit: score on scale] — Range 0-8, higher the score indicates better functioning.
  score on scale | 7.83 (0.4) | 7.91 (0.3) | 7.87 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Completed and Discontinued the Study
Description: Feasibility - Assessment of retention rates.
Time Frame: Baseline to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Mirabegron | Tolterodine Tartrate
Number analyzed (Participants) | 12 | 11
Participants
  Completed study | 11 | 10
  Discontinued Early | 1 | 1
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine Tartrate; Test type: Superiority; p = 0.949, ANCOVA

2. Secondary Outcome: Change From Baseline in California Verbal Learning Test (CVLT) Score at 8 Weeks
Description: Range of 0-80, with the higher the score the better.
Time Frame: Baseline to Week 8
Population: Although 21 participants completed week 8 visits in some form, some participants declined to complete or had missing data for one or more outcome measures at this timepoint.
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Mirabegron | Tolterodine Tartrate
Number analyzed (Participants) | 9 | 8
Score on a Scale | 4.70 [1.13 to 8.27] | 1.59 [-2.20 to 5.37]
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine Tartrate; Test type: Superiority; p = 0.2415, ANCOVA; change from baseline, adjusted for baseline value; Mean Difference (Final Values) = 3.11, 95% CI 2-sided [-2.09 to 8.31]

3. Secondary Outcome: Change From Baseline in Trail Making Test, Trail A Score at 8 Weeks
Description: Trail Making Test, Trail A Time, Range 0-150 seconds, Lower score indicates better functioning
Time Frame: Baseline and 8 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Mirabegron | Tolterodine Tartrate
Number analyzed (Participants) | 10 | 9
seconds | -11.34 [-15.57 to -7.11] | 0.67 [-3.79 to 5.13]
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine Tartrate; Test type: Superiority; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -12.01, 95% CI 2-sided [-18.16 to -5.87]

4. Secondary Outcome: Change From Baseline in Short Physical Performance Battery (SPPB) Score at 8 Weeks
Description: Physical function/mobility, Range 0-12, the higher the score the better.
Time Frame: Baseline to Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mirabegron | Tolterodine Tartrate
Number analyzed (Participants) | 10 | 8
score on a scale | -0.39 [-1.03 to 0.25] | 0.24 [-0.47 to 0.96]
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine Tartrate; Test type: Superiority; p = 0.1956, ANCOVA; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.59 to 0.33]

5. Secondary Outcome: Change From Baseline in Total Urinary Incontinence Frequency Measured by a Voiding Diary at 8 Weeks
Description: Study participants record number of urinary incontinence episodes in a voiding diary. The total urinary incontinence frequency is the sum of urinary incontinence episodes per day.
Time Frame: Baseline to Week 8
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: episodes per day
Arm/Group | Mirabegron | Tolterodine Tartrate
Number analyzed (Participants) | 10 | 9
episodes per day | -2.04 [-3.10 to -0.99] | -3.91 [-5.02 to -2.80]
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine Tartrate; Test type: Superiority; p = 0.0168, ANCOVA; Mean Difference (Final Values) = 1.87, 95% CI 2-sided [0.34 to 3.40]

6. Secondary Outcome: Change From Baseline in Urge Incontinence Episodes Per Day on a Voiding Diary at 8 Weeks.
Description: The sum of urge type incontinence episodes reported by participants on a voiding diary per day.
Time Frame: Baseline and 8 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: episodes per day
Arm/Group | Mirabegron | Tolterodine Tartrate
Number analyzed (Participants) | 10 | 9
episodes per day | -1.64 [-2.73 to -0.54] | -3.74 [-4.90 to -2.58]
Statistical Analysis 1: Comparison: Mirabegron vs Tolterodine Tartrate; Test type: Superiority; p = 0.0101, ANCOVA; Mean Difference (Final Values) = 2.10, 95% CI 2-sided [0.50 to 3.71]

ADVERSE EVENTS:
Time Frame: Baseline to Week 8
Arm/Group | Mirabegron | Tolterodine Tartrate
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 5/12 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron (N=12) | Tolterodine Tartrate (N=11)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cold/flu (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry mouth (General disorders) | 0 (0) | 3 (3)
Memory problems/confusion (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stye (Eye disorders) | 1 (1) | 1 (1)
Blurry vision (Eye disorders) | 0 (0) | 1 (1)
Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Frequent urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Drowsy (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02436889/Prot_SAP_000.pdf